CLINICAL TRIAL: NCT03187730
Title: Integrating Financial Management Counseling and Smoking Cessation Counseling to Reduce Health and Economic Disparities in Low-Income Immigrants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16-02177
Record Dates: First submitted 2017-06-08; First posted 2017-06-15 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Smoking Cessation
Keywords: Smoking Cassation; Immigrants; Economic Disparity
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Active Comparator)
  Interventions: Behavioral: Integrated Smoking Cessation and Financial Counseling; Drug: Nicotine Replacement Therapy (NRT)
- Waitlist Control (Placebo Comparator)
  Interventions: Behavioral: Waitlist Integrated Smoking Cessation and Financial Counseling; Drug: Nicotine Replacement Therapy (NRT)

INTERVENTIONS:
Behavioral: Integrated Smoking Cessation and Financial Counseling — Participants in the intervention group will receive up to nine counseling sessions that integrate two evidence-based counseling approaches: financial management counseling and smoking cessation counseling. Participants will also be eligible to receive a free four-week supply of NRT. Participants will be surveyed at baseline, 2- months, 6-months and 12-months to assess outcomes and treatment satisfaction.
  Arms: Intervention Arm
Behavioral: Waitlist Integrated Smoking Cessation and Financial Counseling — Control participants in the waitlist control group will receive usual care for the first 6 months of the study, while the Intervention Arm receives integrated counseling. The waitlist control group will receive the same counseling program as the Intervention group 6 months after enrollment (up to nine counseling sessions and four weeks of NRT). Participants will be surveyed at baseline, 2-months, 6-months and 12-months to assess outcomes and treatment satisfaction.
  Arms: Waitlist Control
Drug: Nicotine Replacement Therapy (NRT) — Participants in both arms will be eligible to receive a free four-week supply of NRT.

SUMMARY:
This is a 24 month pilot project that will implement and evaluate an innovative program that integrates financial counseling with smoking cessation counseling for low-income immigrants.

DETAILED DESCRIPTION:
This is a two-arm randomized, wait-list control study with 610 participants total: 600 patient participants and 10 staff participants. 600 smokers will be recruited to complete a 9-week intervention that integrates financial management and smoking cessation counseling. Participants will be randomized (300 per arm, stratified by site) to receive the intervention immediately after enrolling (Intervention Arm) or 6 months later (Waitlist Control Arm). Both arms will receive nicotine replacement therapy (NRT) for four weeks as part of their time in integrative counseling. Participants will be observed at baseline, 2 months, 6 months and 12 months to assess outcomes and their satisfaction with treatment.

ELIGIBILITY:
Inclusion Criteria:

* Smokes ≥5 cigarettes per day
* Born outside the U.S.
* Interested in receiving smoking and financial counseling
* Self-reported income below 200% of the current federal poverty level for a given household composition
* New York City resident
* English or Spanish language
* Able to provide informed consent, and
* Does not have a representative who manages his/her funds (to ensure the participant has the ability to manage household money). We will exclude participants who report being pregnant or breastfeeding (unable to receive NRT).

Hospital staff participants:

* Must be current medical or non-medical provider or administrator at Bellevue Hospital or New York University Lutheran Medical Center

Exclusion Criteria:

* We will exclude participants who report being pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Rogers, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Rogers ES, Wysota CN, Sherman SE. Banking Status as a Moderator of Outcomes in a Randomized Controlled Trial Targeting Financial Stress and Smoking. J Gen Intern Med. 2025 Dec 2. doi: 10.1007/s11606-025-10064-0. Online ahead of print. PMID 41331201
- [Derived] Tempchin J, Vargas E, Sherman S, Rogers E. Predictors of Counseling Participation Among Low-Income People Offered an Integrated Intervention Targeting Financial Distress and Tobacco Use. Prev Sci. 2023 Apr;24(3):525-534. doi: 10.1007/s11121-022-01416-x. Epub 2022 Aug 6. PMID 35932394
- [Derived] Rogers ES, Rosen MI, Elbel B, Wang B, Kyanko K, Vargas E, Wysota CN, Sherman SE. Integrating Financial Coaching and Referrals into a Smoking Cessation Program for Low-income Smokers: a Randomized Waitlist Control Trial. J Gen Intern Med. 2022 Sep;37(12):2973-2981. doi: 10.1007/s11606-021-07209-2. Epub 2022 Jan 11. PMID 35018561

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm | Waitlist Control
Started | 208 | 202
Completed | 129 | 154
Not Completed | 79 | 48

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Waitlist Control | Total
Number analyzed (Participants) | 208 | 202 | 410
Age, Continuous [Mean (Full Range); unit: years] | 53.2 [19 to 81] | 52.5 [21 to 78] | 52.85 [19 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 77 | 146
  Male | 139 | 125 | 264
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 105 | 117 | 222
  Not Hispanic or Latino | 103 | 85 | 188
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 9 | 15
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 98 | 92 | 190
  White | 42 | 39 | 81
  More than one race | 7 | 16 | 23
  Unknown or Not Reported | 51 | 43 | 94
Region of Enrollment [Number; unit: participants]
  United States | 208 | 202 | 410

OUTCOME MEASURES:

1. Primary Outcome: % of Participants Who Had Smoked Cigarette(s) in the Past 7 Days (at 6 Months From Baseline)
Description: Participants answered "In the past 7 days, have you smoked a cigarette? (yes/no)"; % of "yes" is reported per arm
Time Frame: 6 Months
Measure: Number; unit: % of participants
Arm/Group | Intervention Arm | Waitlist Control
Number analyzed (Participants) | 128 | 155
% of participants | 27 | 13

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intervention Arm | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 3/208 | 1/202
Serious Adverse Events (participants affected / at risk) | 11/208 | 5/202
Other Adverse Events (participants affected / at risk) | 0/208 | 0/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=208) | Waitlist Control (N=202)
Hospitaliztion (General disorders) | 11 (11) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT03187730/Prot_SAP_000.pdf